CLINICAL TRIAL: NCT02903108
Title: Clinical Efficacy of Subgingivally Delivered 0.75% Boric Acid Gel As An Adjunct to Mechanotherapy in Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Clinical Efficacy of 0.75% Boric Acid Gel in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014O
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Boric acid group (Active Comparator): Oral prophylaxis followed by 0.75% boric acid drug in gel form placed in intrabony defects
  Interventions: Drug: SRP plus boric acid gel
- Placebo group (Placebo Comparator): Oral prophylaxis followed by placebo gel placement in intrabony defects
  Interventions: Drug: SRP plus placebo gel

INTERVENTIONS:
Drug: SRP plus boric acid gel — SRP followed by 0.75% boric acid placement into intrabony defect
  Arms: Boric acid group
Drug: SRP plus placebo gel — SRP followed by placebo gel placement into intrabony defect
  Arms: Placebo group

SUMMARY:
The purpose of the present study was to evaluate the effects of subgingival delivery of boric acid gel as an adjunct to scaling and root planing in chronic periodontitis (CP) patients.

DETAILED DESCRIPTION:
Background: The purpose of this double-masked, randomized, controlled clinical trial was to evaluate the effects of subgingival delivery of boric acid gel as an adjunct to scaling and root planing (SRP) on clinical and radiographic parameters and compare this method with SRP plus placebo gel alone in with chronic periodontitis (CP) patients.

Methods: Thirty nine systemically healthy patients with CP are included in this study. They were divided into two groups: 1) SRP + 0.75% Boric acid gel (BA group); 2) SRP + Placebo gel (Placebo group). At baseline, 3 month, and 6 months after treatment, clinical measurements, including plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), clinical attachment level (CAL) and radiographic parameters intrabony defect depth (IBD), percentage change in radiographic defect depth reduction (DDR%) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy with deep pockets (PD of ≥5mm or CAL ≥4mm) and vertical bone loss ≥3 mm on intraoral periapical radiographs
* Patients with ≥20 teeth with no history of periodontal therapy in the preceding 6 months nor under any antibiotic therapy

Exclusion Criteria:

* Patients on systemic boron therapy
* Known or suspected allergy to boron supplementation
* Patients with aggressive periodontitis
* Tobacco use in any form, smokers, alcoholics
* Immunocompromised and systemically unhealthy patients
* Pregnant or lactating females

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Defect depth reduction (%) | Change from baseline to 6 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth (mm) | Change from baseline to 6 months
  measured in mm
clinical attachment level (mm) | Change from baseline to 6 months
  measured in mm
modified sulcus bleeding index | Change from baseline to 6 months
  scale from 0-3
plaque index | Change from baseline to 6 months
  scale from 0-3

CONTACTS AND LOCATIONS:
Locations (1):
- Bangalore, Karnataka, India